CLINICAL TRIAL: NCT06850376
Title: COVID Feel Good-An Easy Self-Help Virtual Reality Protocol to Overcome the Psychological Burden of Coronavirus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: Clemson University (Virtual Reality and Nature Lab) (Unknown); University of Barcelona (Other); University of Tsukuba (Other); Konkuk University (Other); University of Bergen (Other); University of Liege (Other); Catholic University of the Sacred Heart (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 39C001
Record Dates: First submitted 2025-02-26; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: COVID-19 Pandemic Psychological Impact; Stress; Anxiety Disorders; Depression; Social Isolation
Keywords: Virtual Reality; Self-help Mental Health; Relaxation; Social Connectedness; Pandemic Coping; Nature; Simulation
MeSH Terms: conditions — Anxiety Disorders; Depression; Social Isolation

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either an experimental group receiving the 7-day VR self-help protocol immediately, or a waiting-list control group that receives the intervention after the initial waiting period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR Self-Help Protocol (Experimental): Participants in this arm receive the 7-day COVID Feel Good self-help protocol immediately upon enrollment. The intervention consists of daily exposure to the 'Secret Garden' 360° VR video combined with specific daily cognitive and social exercises. Participants use a VR headset compatible with the Cardboard format to experience the 10-minute VR video once per day for 7 consecutive days, followed by completing the daily exercise with a partner.
  Interventions: Behavioral: COVID Feel Good VR Self-Help Protocol
- Waiting List Control (Other): Participants in this arm are placed on a waiting list for 7 days before receiving the intervention. During this waiting period, they complete the same baseline assessments as the experimental group but do not receive any specific intervention. After the 7-day waiting period, these participants then receive the same 7-day VR self-help protocol.
  Interventions: Other: Waiting Period

INTERVENTIONS:
Behavioral: COVID Feel Good VR Self-Help Protocol — The intervention consists of a 7-day self-help protocol based on daily exposure to 'The Secret Garden' 360° VR video (10 minutes per day) available at www.covidfeelgood.com, combined with different daily cognitive and social exercises. Participants use a smartphone with VR headset compatible with the Cardboard format. Each day's exercise addresses different psychological aspects: fighting rumination, awakening self-esteem, autobiographical memory, sense of community, goals and dreams, empathy, and planning for change. Exercises are designed to be performed individually and then discussed with a partner.
  Arms: VR Self-Help Protocol
Other: Waiting Period — Participants in the control group initially undergo a 7-day waiting period before receiving the VR self-help protocol. During this period, they complete the same baseline assessments as the experimental group but do not receive any specific intervention.
  Arms: Waiting List Control

SUMMARY:
This pragmatic trial aims to evaluate whether a weekly self-help virtual reality protocol can help overcome the psychological burden of the COVID-19 pandemic. The protocol is based on 'The Secret Garden' 360° VR video available online (www.covidfeelgood.com) which simulates a natural environment to promote relaxation and self-reflection. The VR experience is combined with daily cognitive and social exercises designed to facilitate critical examination of personal identity, relationships, and coping strategies. The study assesses whether this intervention can reduce anxiety, depression, perceived stress, and hopelessness while improving well-being and social connectedness during pandemic-related restrictions.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants (≥18 years)
* Native speakers of the country where they will be enrolled
* Have experienced at least two months of quarantine or isolation related to the coronavirus pandemic
* Provide full, written, informed consent
* Have the availability of a smartphone and a cardboard VR headset
* Availability and agreement of a partner for conducting the self-help component of the treatment

Exclusion Criteria:

* Visual or hearing impairments that can limit the participation in the protocol
* Participants reporting vestibular and/or balance disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in depression, anxiety, and stress levels as measured by Depression Anxiety Stress Scale (DASS-21) | Baseline (Day -7 and Day 0), Post-intervention (Day 7), and 2-week Follow-up (Day 21)
  The Depression Anxiety Stress Scale (DASS-21) is a self-report questionnaire consisting of 21 items divided into three subscales that measure depression, anxiety, and perceived stress. Each subscale can be computed individually or added together into a score for general distress. Higher scores indicate greater symptoms of depression, anxiety, and stress. The scale will be used to assess changes in psychological distress associated with the COVID-19 pandemic before and after the VR self-help intervention.
Perceived Stress Scale (PSS-10) | Baseline (Day -7 and Day 0), Post-intervention (Day 7), and Follow-up (Day 21)
  A scale measuring subjective perception of stress during the past week
Change in hopelessness levels | Baseline (Day -7 and Day 0), Post-intervention (Day 7), and Follow-up (Day 21)
  A scale measuring pessimistic attitudes toward the future

SECONDARY OUTCOMES:
Change in social connectedness | Baseline (Day -7 and Day 0), Post-intervention (Day 7), and 2-week Follow-up (Day 21)
  A scale measuring sense of connection to others and to the social context
Change in fear of coronavirus | Baseline (Day -7 and Day 0), Post-intervention (Day 7), and Follow-up (Day 21)
  A scale measuring level of fear related to the COVID-19 pandemic
Change in relaxation levels during intervention | Daily during intervention (Days 1-7)
  A scale measuring relaxation and perceived stress during the intervention
Change in subjective distress during intervention | Daily during intervention (Days 1-7)
  A scale measuring level of perceived distress

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Auxologico Italiano, Milan, Lombardy, Italy